CLINICAL TRIAL: NCT06899750
Title: E3 Hypertension - A Team-based, Multidisciplinary Model in Addressing Barriers to Hypertension Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24100803
Record Dates: First submitted 2025-03-11; First posted 2025-03-28 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Hypertension
Keywords: hypertension; self-monitoring; social determinants of health; adherence
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertension Team Based Group (Experimental): A multidisciplinary team composed of a pharmacist, social worker, and nurse coupled to a self-monitoring blood pressure phone app will provide hypertension monitoring, medication titration, diet and lifestyle education, and referrals for social needs. The team will interact with the patients predominantly via tele-health remotely for 6 months.
  Interventions: Behavioral: E3 Multidisciplinary Team
- Hypertension Self-Guided Group (Active Comparator): A research assistant ensures patients in the self-guided group have a home blood pressure monitor on enrollment and will call patients at 3 and 6 months to ensure the blood pressure monitor is functioning correctly and to remind patients to check their blood pressure and follow-up with their primary care doctors. Patients will continue with standard clinical care for hypertension in addition to receiving timed, mailed educational materials on hypertension, remote monitoring, diet and lifestyle recommendations for 6 months.
  Interventions: Behavioral: E3 Self-Guided Hypertension Education Program

INTERVENTIONS:
Behavioral: E3 Multidisciplinary Team — The E3 Multidisciplinary team is composed of a remote pharmacist, social worker, and nurse working together with patients via a remote monitoring, educational hypertension phone app to overcome barriers to hypertension control via behavioral change, medication adherence and titration, diet and lifestyle education and resource referrals for social needs.
  Arms: Hypertension Team Based Group
Behavioral: E3 Self-Guided Hypertension Education Program — Patients will receive timed, mailed educational materials on hypertension self-monitoring, diet and lifestyle modifications to supplement usual clinic-based hypertension care with their primary care doctor. A research assistant will ensure patients have home blood pressure monitors on enrollment, and will remind patients to check their blood pressures and follow-up with their primary care doctors at 3 months and 6 months.
  Arms: Hypertension Self-Guided Group

SUMMARY:
This study aims to compare a multidisciplinary clinical hypertension and social needs intervention to enhanced standard of care for hypertension management in primary care clinics with regards to hypertension control outcomes.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death in the US as well as in Chicago. Risk factors for CVD include hypertension, diabetes, and lifestyle factors such as smoking, diet, and obesity. Among the critical social and structural determinants of cardiovascular health are food access, neighborhood safety, education, poverty, and chronic stress. Chicago and its surrounding region suffer from longstanding racial disparities in both social conditions and chronic disease burden, contributing to stark racial gaps in cardiometabolic disease mortality. Life expectancy is as high as 84 years on Chicago's North Side, but only 68 years on the West Side - a gap of 16 years.

Rush has collaborated with Novartis to "close the gap" in CVD inequities on Chicago's West Side by concentrating a critical mass of resources on community-centric approaches to wellness, prevention and management. Engage, Empower, Evaluate (E3) has been built on the foundation of Rush's mission to ensure that all patients and individuals at risk of developing CVD on Chicago's West Side receive the care they need, regardless of race/ethnicity, socioeconomic status, gender, or neighborhood, with the ultimate goal to reduce the CVD life expectancy gap for West Side residents by 50% by 2030. To do so, the study team coordinated clinical and community programming into a seamless health-promoting environment, tailored to the specific needs of the population, through remote monitoring and a multidisciplinary team composed of a nurse, social worker, and pharmacist.

The study team now proposes a trial of the E3 intervention, a remote hypertension monitoring, social care, medication adherence and behavioral lifestyle intervention to improve hypertension control among African American and Latinx patients attending primary care clinics at Rush University Medical Group locations with the eventual aim of closing the racial/ethnic disparity in hypertension control. The proposed feasibility trial will use a randomized-control, four-pronged approach to improve hypertension control. The intervention group will receive the following: 1) remote blood pressure monitoring, 2) a multidisciplinary team composed of nurse, pharmacist and social worker to address medical and social needs, 3) medication titration and adherence support, and 4) a culturally tailored hypertension self-management and diet education mobile phone application. The control group will receive an enhanced version of standard of care for hypertension through a home blood pressure cuff, and dietary and lifestyle educational materials tailored to hypertension self-management sent at timed intervals. The study team hypothesizes that the E3 Hypertension program participants will achieve a greater decrease in systolic blood pressure, and a greater percentage will have reduction of blood pressure below stage 2 hypertension (<140/90) in comparison to the control group receiving enhanced standard of care for hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* African American and/or Latinx
* Uncontrolled stage 2 hypertension, BP >/= 140/90
* Patient is following with Rush primary care provider in eligible Rush primary care clinics
* Patient has a smart phone (Android or iOS)
* Patient has an email

Exclusion Criteria:

* Organ transplant recipient
* On dialysis
* Patient is already participating in another remote hypertension monitoring program
* Patient is not interested in participating in the program
* Patient has already participated in the E3 Hypertension program or the E3 Diabetes program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure change at 6 months | 6 months
  Percentage of participants with a decrease in systolic blood pressure of at least 10mmHg between pre and post clinic-based blood pressure measurements.

SECONDARY OUTCOMES:
Hypertension control at 9 months | 9 months
  Percentage of participants with hypertension control (BP< 140/90) at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Pallok, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared, however aggregate patient data may be shared with other researchers

DOCUMENTS (1):
  • Informed Consent Form (2025-03-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT06899750/ICF_000.pdf